CLINICAL TRIAL: NCT05454605
Title: Оptical Spectroscopy in the Diagnosis of Intra-articular Injuries of the Knee Joint
Brief Title: Оptical Spectroscopy in the Diagnosis of Intra-articular Injuries
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 01-22
Record Dates: First submitted 2022-05-12; First posted 2022-07-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-05

CONDITIONS: Cartilage Destruction
Keywords: cartilage; regeneration; destruction; knee; intraarticular lesions

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1, ex vivo: 1. Assessment of the degree of cartilage damage according to the International Cartilage Regeneration & Joint Preservation Society (ICRS) classification.
  2. Optical spectroscopy of patient tissue samples.
  3. Study of the mechanical properties of intra-articular tissues and cartilage thickness with an indenter.
  4. Histological assessment of tissues according to the Osteoarthritis Research Society International (OARSI) classification.
- group 2, in vivo: 1. Assessment of the degree of cartilage damage according to the ICRS classification.
  2. Optical spectroscopy during arthroscopy/arthroplasty.
  3. Magnetic resonance imaging (MRI).

SUMMARY:
Intra-articular joint injuries are the most common and prognostically unfavorable in case of untimely or erroneous diagnosis, which leads to a significant violation of the quality of life and activity of patients. For example, untimely diagnosis and determination of the degree of damage to the subchondral bone can lead to progression, namely, an increase in the edema zone with transformation into an irreversible process - avascular necrosis of the bone. Mistakes in diagnosing subsynovial injuries of the ligamentous apparatus and assessing its functional viability can lead to the development of chronic joint instability, chronic synovitis, and progression of intraarticular destruction.

Methods of early and accurate diagnosis allow timely and personalized treatment, they are aimed at preventing the development of complications and the need for repeated expensive and often disabling operations. The issue of developing the method of intraoperative navigation with the use of quantitative assessment methods in operations on the musculoskeletal system is also relevant.

In this regard, the methods of optical spectroscopy and optoacoustics proposed in the project, which can solve the above problems, are of particular relevance.

Thus, the scientific problem to be solved by the proposed project is the development of optical and optoacoustic spectroscopy methods for biomedical diagnostics. The development of new methods and tools capable of detecting and characterizing both early and hidden predictors of the possible progression of osteoarthritis will prevent or reduce the risks of possible complications and irreversible intra-articular changes.

DETAILED DESCRIPTION:
The objectives of this work is to create new optical methods for in vivo analysis of the state of cartilage tissue.

Methods: A prospective study will develop an instrument that implements two optical methods for assessing the condition of cartilage tissue: diffuse reflectance spectroscopy (DRS) and near-infrared fluorescence spectroscopy. Explants (knee joint) will be used as experimental material. To assess the diagnostic capabilities of optical spectroscopy methods, studies of the mechanical characteristics of cartilage will be carried out simultaneously with the optical characteristics. Cartilage mechanical parameters will be measured using a Mach-1 v500c indenter (Biomomentum, Laval, QC, Canada) equipped with a three-axis dynamometer. The direction of the normal to the sample will be measured with a spherical indenter; a needle puncture will be performed to assess the thickness of the explant tissue. Measurements will determine the Young's modulus, the direction of the normal and the thickness of the cartilage. This work is supported by the Russian Science Foundation (grant no. 21-79-10325).

An indentation will be performed to determine the mechanical parameters of the cartilage at different points and to obtain DCR spectra of the cartilage in the wavelength range of 850-1050 nm.Analysis of changes in the properties of water in the cartilaginous tissue of the knee joint in normal and pathological conditions will be supplemented by a study of its own IR fluorescence. In preliminary experiments, it was found that different parts of the cartilage of different explants have different levels of red fluorescence at different stages of degeneration, however, in order to draw conclusions, it is necessary to expand the number of measured samples to assess the reliability of the results of the observed differences.

In the course of the work, a mobile unit will be developed that implements the methods of fluorescence spectroscopy in the near infrared range and DLS, and the mechanical properties of explants will also be studied. In the future, it is planned to use the developed technique for assessing the state of the cartilage intraoperatively.

Before conducting the experimental work, it is planned to write a systematic review on the research topic.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of the patient to participate in the study.
2. The age of the patient is from 18 to 85 years.
3. Gender male and female.
4. The patient has intra-articular injuries of the knee joint.

Exclusion Criteria:

1. Refusal to participate in the study and to sign informed consent.
2. The age of the patient is less than 18 and more than 85 years.
3. Pregnancy, lactation.
4. The presence of severe concomitant somatic pathology (diseases of the cardiovascular system, lungs, liver and kidneys), decompensated diabetes mellitus.
5. Oncological diseases.
6. Mental illness.
7. Alcohol abuse or drug use.
8. Chronic viral and bacterial infections in the acute stage.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Work will be carried out with biological samples of bone and cartilage tissue in compliance with all ethical standards: work with explants (38 samples), as well as in vivo measurements - intraoperatively (10 patients).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Measurement of mechanical properties and application of cartilage by indentation method | The processing of the received data will be carried out from March 2022 to December 2023.
  Micromechanical system Mach-1™ v500csst (Biomomentum Inc., Laval, Quebec, Canada) allows to perform normal alignment and indentation mapping by simultaneously moving the three stages with the use of multiple-axis load cell. After mapping in the normal indentation mode, the cartilage thickness was measured at the same points in the mapping mode by needle penetration technique.
  The Lee-Radock model corrected for the finite local thickness of the soft layer was used to estimate the mechanical parameters. The experimental curves were processed by the standard Hertz's model. Numerical processing was performed in MATLAB (MathWorks, USA) using previously developed algorithms.
  A standard linear solid (SLS) model was chosen as a relaxation function to describe experiments on indentation-relaxation tests of cartilage tissue, where the main parameters are: instantaneous Young modulus E0, equilibrium Young modulus E, and relaxation time.
Reflectance and Cartilage Water Measurement by Diffuse Reflectance Spectroscopy (DRS) | The processing of the received data will be carried out from March 2022 to December 2023.
  DRS measurements were performed in the spectral region of 850-1050 nm. The tungsten-halogen lamp (Thorlabs, Germany) was used as a light source. The measurements were performed with two 550 μm fibers with a 2.5 mm distance between the centers of their faces, the first one guiding the light to the sample and the second one attached to the QE65000 spectrometer (OceanOptics, USA). For spectra measurement, a specially probe was used, which makes it possible to use it in conjunction with the micromechanical tester setup.
  Before each series of experiments, the reference spectrum (reflection from the reference diffuse reflectance) and the background spectrum are measured, and the reflectance and effective optical density are calculated.
Simulation of light propagation in the explant by the Monte Carlo method. | The processing of the received data will be carried out from March 2022 to December 2023.
  In order to estimate the dependencies of the observed parameters on the properties of tissue such as cartilage thickness, water content and scattering properties, light propagation in the explant was simulated using the Monte Carlo method. The explant was modeled as a medium consisting of 2 distinct layers with individual scattering and absorption properties. The first layer represented cartilage, where the main absorption is determined by the OH line of water at ~980 nm, the second layer represented bone tissue, whose absorption possesses a local maximum at ~930 nm, determined by the CH line of the bone matrix.
Assessment of the comparison of osteoarthritis grades according to ICRS using the nonparametric Mann-Whitney U-test | The processing of the received data will be carried out from March 2022 to December 2023.
  Multiple-group statistical comparisons among different ICRS osteoarthritic grades were assessed by nonparametric Mann-Whitney U test using custom-made scripts based on the Python programming language with statsmodels, SciPy libraries. In total, 600 DRS spectra obtained for each ICRS grade (i.e., group) of OA cartilage were used for this test. The assumptions (i.e., independent measurements, non-normal distribution, and similar var-iability) of Mann-Whitney U test were verified. The p-values for each pairwise Mann-Whitney U test were then recalculated using the Bonferroni correction. In all multiple-group pairwise comparisons, p-value of less than 0.05 was considered indicative of statistical significance.
Histological examination of bone and cartilage samples | The processing of the received data will be carried out from March 2022 to December 2023.
  For histological examination, samples were fixed in a 10% neutral formalin (HistoSafe, Biovitrum), were decalcified in a special solution (SoftyDek, Biovitrum) during 24 hours, washed in running water for an hour, subjected to standard alcohol wiring and poured with paraffin. 4-μm-thick paraffin sections were stained with Safranin O and fast green according to the standard protocol. The obtained microscopic preparations were studied using a universal microscope LEICA DM4000 B LED (Leica Microsystems, Germany) equipped with a digital video camera LEICA DFC7000 T (Leica Microsystems, Germany). To verify the degree of cartilage degradation, a histological study will carried out on a selection of explants.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Lychagin, Study Chair — IM Sechenov University; Yuliya Goncharuk, Principal Investigator — IM Sechenov University
Locations (1):
- Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No